CLINICAL TRIAL: NCT02630849
Title: Does a Multimodal no-Compression Suture Technique of the Intercostal Space Reduce Chronic Post-Thoracotomy Pain? A Prospective Randomized Study
Brief Title: Does a Multimodal no-Compression Suture Technique of the Intercostal Space Reduce Chronic Post-Thoracotomy Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Mohsen Ibrahim, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1222/13
Record Dates: First submitted 2015-12-07; First posted 2015-12-15 (Estimated); Last update posted 2015-12-15 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- IMF group (Experimental): intercostal muscle flap and pericostal no-compression suture of the intercostal space
  Interventions: Procedure: intercostal muscle flap and pericostal no-compression suture
- IINB group (Active Comparator): Standard suture technique of the intercostal space associated with an intrapleural intercostal nerve block
  Interventions: Procedure: Standard suture technique of the intercostal space

INTERVENTIONS:
Procedure: intercostal muscle flap and pericostal no-compression suture — intercostal muscle flap and pericostal no-compression suture of the intercostal space
  Arms: IMF group
Procedure: Standard suture technique of the intercostal space — Standard suture technique of the intercostal space associated with an intrapleural intercostal nerve block
  Arms: IINB group

SUMMARY:
Chronic post-thoracotomy pain is a significant adverse outcome of thoracic surgery. transcollation technology evaluated with a prospective randomized trial the effect of a multimodal no-compression suture technique of the intercostal space on postoperative pain occurrence in patients undergoing mini-thoracotomy.

Patients undergoing a muscle-sparing lateral mini-thoracotomy for different thoracic diseases were randomly divided into two groups:one group received intercostal muscle flap harvesting and pericostal no-compression "edge" suture (IMF group), and the second group received a standard suture technique associated with an intrapleural intercostal nerve block (IINB group).

The aim of the study was to demonstrate that the multimodal no-compression suture technique is a rapid and feasible procedure reducing early and chronic post-thoracotomy pain intensity.

DETAILED DESCRIPTION:
Patients' data were prospectively recorded in a single database and surgery was performed in a single thoracic center in order to achieve homogenous treatment.

After acceptance from the Ethics Committee of our Institution, a prospective randomized study of 487 patients was performed from October 2011 to October 2013 in the Thoracic Surgery Division - Sant'Andrea Hospital, Faculty of Medicine and Psychology, University of Rome "Sapienza". All patients who were scheduled to undergo a muscle-sparing lateral mini-thoracotomy for different thoracic diseases were eligible for this trial. Exclusion criteria were: history of previous thoracotomy, chronic pain syndrome (any type of pain), opioid/steroid use 6 months before surgery, chest trauma with rib fractures, radiologic evidence of parietal pleural or chest wall tumor invasion, and previous neoadjuvant or radiation therapy.

Preoperative consent was obtained from all patients, informed that they would have one of the two methods of chest closure.

Pulmonary function tests (spirometry and 6-minute walking test [6-MWT]) were performed in all patients preoperatively and at 1 and 6 months postoperatively. All patients received our standard muscle-sparing lateral minithoracotomy through the fifth intercostal space without division of the latissimus dorsi muscle and the serratus anterior muscle. The postoperative analgesic protocol was the same for all patients in both groups, and consisted of a continuous intravenous infusion of tramadol (10 mg/h) and ketorolac tromethamine (3 mg/h), starting at the time of surgical skin incision and continuing until 48-72 h after surgery. Intravenous analgesia was then continued with ketorolac tromethamine (10 mg tid) and paracetamol (1 g tid) until discharge from the hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were scheduled to undergo a muscle-sparing lateral mini-thoracotomy for different thoracic diseases were eligible for this trial.

Exclusion Criteria:

* History of previous thoracotomy
* Chronic pain syndrome (any type of pain)
* Opioid/steroid use 6 months before surgery
* Chest trauma with rib fractures
* Radiologic evidence of parietal pleural or chest wall tumor invasion
* Previous neoadjuvant or radiation therapy.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Long term Brief Pain Inventory Scale Variation | 6 months after surgery
  the aim of the study is to evaluate the variation of the brief pain inventory scale (BPI) in patients treated with a non-divided intercostal muscle flap associated with pericostal "edge" sutures (thus protecting the intercostal nerves from trauma) on long-term versus patients who will receive our standard pain control strategy (intrapleural intercostal nerve block).

SECONDARY OUTCOMES:
Mid term Brief Pain Inventory Scale Variation | 1 month after surgery
  the aim of the study is to evaluate the variation of the brief pain inventory scale (BPI) in patients treated with a non-divided intercostal muscle flap associated with pericostal "edge" sutures (thus protecting the intercostal nerves from trauma) after 1 month versus patients who will receive our standard pain control strategy (intrapleural intercostal nerve block).
Pulmonary functional tests | 6 months after surgery
  spirometry and 6-minute walking test [6-MWT] were evaluated in both groups to assess the differences in lung function

CONTACTS AND LOCATIONS:
Overall Officials: Erino A. Rendina, Professor, Study Chair — University of Roma La Sapienza

REFERENCES:
- [Background] Caraceni A, Mendoza TR, Mencaglia E, Baratella C, Edwards K, Forjaz MJ, Martini C, Serlin RC, de Conno F, Cleeland CS. A validation study of an Italian version of the Brief Pain Inventory (Breve Questionario per la Valutazione del Dolore). Pain. 1996 Apr;65(1):87-92. doi: 10.1016/0304-3959(95)00156-5. PMID 8826494
- [Background] Cerfolio RJ, Bryant AS, Maniscalco LM. A nondivided intercostal muscle flap further reduces pain of thoracotomy: a prospective randomized trial. Ann Thorac Surg. 2008 Jun;85(6):1901-6; discussion 1906-7. doi: 10.1016/j.athoracsur.2008.01.041. PMID 18498792
- [Background] D'Andrilli A, Ibrahim M, Ciccone AM, Venuta F, De Giacomo T, Massullo D, Pinto G, Rendina EA. Intrapleural intercostal nerve block associated with mini-thoracotomy improves pain control after major lung resection. Eur J Cardiothorac Surg. 2006 May;29(5):790-4. doi: 10.1016/j.ejcts.2006.01.002. Epub 2006 Feb 14. PMID 16481188